CLINICAL TRIAL: NCT03729440
Title: Evaluation of Esophageal Injuries in Corrosives in Assiut Governorate - Experimental Comparison Between Different Treatments
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MKMAbdelrahim, assistant lecturer, Assiut University
Other Study IDs: EsophagealCorrosiveAssiut
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Clinico-epidemiological Characteristics of Corrosive Patients Presenting at Assiut Governorate
MeSH Terms: interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- corrosive patients
  Interventions: Behavioral: development of complications or not

INTERVENTIONS:
Behavioral: development of complications or not — assessment of development of complications

SUMMARY:
Esophageal stricture is one of the most common sequelae of caustic injury. Up to 70% of patients with grade IIB and more than 90% of patients with grade III injury are likely to develop esophageal stricture. Stricture formation can be prevented by suppressing fibrosis and scar formation therefore; many agents are explored for treatment on various models in this subject.

DETAILED DESCRIPTION:
In spite of the multiple efforts to educate the public, Caustic ingestion maintains its place as an important public health issue due to the availability of caustic agents and the loose regulatory control on its production. All the cases will be evaluated by detailed history and thorough physical examination and necessary investigations. Patient's sheet will include; name, age, sex, occupation, residence, type of administrated substance, route and mode of exposure, symptoms and sighs (pain , vomiting , diarrhea) and any received treatment.

ELIGIBILITY:
Inclusion Criteria:

-1- All the cases with the primary diagnosis of acute caustic injury will be included in the study.

2- Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

* 1- Caustic substance ingested patient with any chronic disease. 2- Patients with history of congenital esophageal stricture. 3- Unable to provide informed consent. 4- Unlikely to return at 8 weeks. 5- Ingestion of substances other than corrosive (co-ingestion).

Ages: 6 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cases diagnosed as acute corrosive toxicity which admitted to emergency unit Assiut University Hospital ,children university hospital and ministry of health hospitals in Assiut in duration of one year.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
fate of cases | 6 months
  development of esophageal stricture or not